CLINICAL TRIAL: NCT02286362
Title: An Observational Study of the Safety of Herceptin Given Subcutaneously in Patients With Early HER2-positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28983
Record Dates: First submitted 2014-10-30; First posted 2014-11-07 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This non-interventional prospective study will assess the safety of Herceptin SC (subcutaneous administration) as used in routine clinical practice. Patients with HER2-positive early breast cancer, naive and non-naive of HER2+ treatment who are to be treated in the neoadjuvant and adjuvant setting and scheduled to initiate a treatment with Herceptin SC in routine clinical practice use are eligible to participate. The total study duration is anticipated to be 38 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged >/= 18 years
* Patients with HER2-positive early breast cancer who according to national guidelines are eligible for neoadjuvant or adjuvant HER2+ treatment
* Patients for whom the investigator has decided to start a treatment with Herceptin SC
* Trastuzumab treatment naive or non-naive (previously intravenous treatment)
* Informed consent

Exclusion Criteria:

* Patients previously treated with Herceptin SC treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive early breast cancer scheduled to initiate a treatment with Herceptin SC.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Safety (composite outcome measure): Incidence, nature, and severity according to NCI-CTCAE v. 4.0 of: adverse events (AEs), serious AEs, grade >/= 3 AEs, non-serious adverse drug reaction or causality unknown, AESI (congestive heart failure) | approximately 13 months

SECONDARY OUTCOMES:
Demographic data | Up to 12 months
Number of modalities regarding dose and injection site of Herceptin SC administration | Up to 12 months
Patient-reported outcome: Quality of Life using the EORTC QLQ-C30 questionnaire | Every 3 months, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (97):
- France (97):
  - Clinique Du Docteur Calabet; Cromg, Agen
  - C H Du Pays D'Aix En Provence; Hopital De Jour, Aix-en-Provence
  - Ch Du Pays D Aix; Maternite Gynecologie, Aix-en-Provence
  - Poly Parc Rambot La Provencale; Chimiotherapie Ambulatoire, Aix-en-Provence
  - Centre Hospitalier Albi; Oncologie, Albi
  - Clinique Claude Bernard; Onco Hematologie, Albi
  - Hopital Prive D Antony; Oncologie, Antony
  - Cmc De Tronquieres;Chimiotherapie Et Radiotherapie, Aurillac
  - Ch D Auxerre; Oncologie, Auxerre
  - Clinique Du Docteur Maymard; Hopital De Jour Chimiotherapie, Bastia
  - Hopital De Falconaja Furiani; Hopital De Jour, Bastia
  - Centre Oncologie Du Pays Basque, Bayonne
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Centre Pierre Curie, Beuvry
  - Ch De Beziers; Hematologie, Béziers
  - Hopital Avicenne; Cancerologie, Bobigny
  - Clinique Tivoli; Chimiotherapie Radiotherapie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Clinique Pasteur Lanroze; Chimiotherapie Radiotherapie, Brest
  - CMC de Bligny; Oncologie Court Sejour, Briis-sous-Forges
  - Hopital Pierre Nouveau; Medecine A, Cannes
  - CH Carcassonne; Service Onco Hematologie, Carcassonne
  - Clinique Montreal; Chimiotherapie, Carcassonne
  - Medipole De Savoie; Departement Oncologie, Challes-les-Eaux
  - Hopital Prive Paul d Egine; Chimiotherapie Ambulatoire, Champigny-sur-Marne
  - CH de Cholet; oncologie, Cholet
  - Hopital Antoine Beclere; Hopital De Jour, Clamart
  - Centre De Radiotherapie Et D'Oncologie; Oncologie, Compiègne
  - Groupe Hospitalier Public Du Sud De L'Oise GHPSO; Oncologie, Creil
  - Chi De Creteil; Radiotherapie Oncologie, Créteil
  - Hopital Henri Mondor; Oncologie Medicale, Créteil
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Centre De Radiotherapie Du Parc, Dijon
  - Ch De La Dracenie; Hopital De Jour, Draguignan
  - Clinique Claude Bernard; Chimiotherapie, Ermont
  - Chi Emile Durkheim Site Epinal; Oncologie, Épinal
  - Chi De Frejus Saint Raphael; Oncologie, Fréjus
  - Chi Alpes Du Sud Site De Gap; Med Interne Et Polyvalente, Gap
  - Centre Mistral; Chirurgie Cancerologie Gynecologiques, Guilherand-Granges
  - CH de Marne la vallee; Oncologie Medicale, Jossigny
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Hopital Louis Pasteur; Oncologie Hematologie, Le Coudray
  - Ch Du Mans; Medecine Hematologie Oncologie, Le Mans
  - Polyclinique Du Bois; Oncologie, Lille
  - Clinique Chenieux; Oncology, Limoges
  - Ch De Longjumeau; Hopital De Jour Et Semaine, Longjumeau
  - Ch De Lons Le Saunier; Medecine 5, Lons-le-Saunier
  - Ch Bretagne Sud Site Scorff; Oncologie Medicale, Lorient
  - Clinique De La Sauvegarde; Chimiotherapie, Lyon
  - Clinique Saint Faron; Sce Oncologie Radiotherapie, Mareuil-lès-Meaux
  - Ctre Hosp Prive Beauregard; Hop De Jour Chimiotherapie, Marseille
  - Hopital Clinique Claude Bernard; Oncologie Medicale, Metz
  - Hopital Layne; Medecine Ambulatoire, Mont-de-Marsan
  - Ghi Le Raincy Montfermeil; Oncologie Medicale, Montfermeil
  - Ch De Montlucon; Hematologie Cancerologie, Montluçon
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Centre Catherine de Sienne; Chimiotherapie, Nantes
  - Polyclinique Du Languedoc; Chimiotherapie, Narbonne
  - Ch Georges Renon; Oncologie Radiotherapie, Niort
  - Hopital Caremeau; Hematologie Oncologie, Nîmes
  - Hopital Caremeau; Maternite Gynecologie, Nîmes
  - Clinique Valdegour, Nîmes
  - CROM, Osny
  - Ch Pitie Salpetriere; Oncologie Medicale, Paris
  - GH Paris Saint Joseph; Hopital De Jour Oncologie, Paris
  - Ch Francois Mitterrand; Medecine Oncologie, Pau
  - Centre Catalan D' Oncologie, Perpignan
  - Hopital Saint Jean; Centre Henri Pujol, Perpignan
  - Polyclinique Francheville; Med Chimiotherapie Radiotherapie, Périgueux
  - CH Rene Dubos; Oncologie, Pontoise
  - CH Annecy Genevois site Annecy; Oncologie, Pringy
  - Chi De Cornouaille; Oncologie Hospitalisation, Quimper
  - Institut Jean Godinot; Pavillon Rubis, Reims
  - Clinique de la Theuillerie; Oncologie, Ris-Orangis
  - Clinique Armoricaine Radiologie; Cons Externes, Saint-Brieuc
  - Clinique Francois 1er; Service De Chimiotherapie, Saint-Dizier
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Clinique de L'Union; Oncologie, Saint-Jean
  - CH de Saint Jean De Maurienne; Had St Jean De Maurienne, Saint-Jean-de-Maurienne
  - Clinique Mutualiste L Estuaire, Saint-Nazaire
  - Centre Hospitalier De Sens; Medecine Generale Oncologie, Sens
  - Ch Gaston Ramon; Hopital De Jour, Sens
  - Centre Clinical; Oncologie Medicale, Soyaux
  - Clinique De L Estree; Oncologie Medicale, Stains
  - Clinique Medico Chir Charcot; Chir Cancerologie, Ste Foy Les Lyon
  - Institut D Oncologie Medical, Strasbourg
  - Strasbourg Oncologie Libérale, Strasbourg
  - Hopital Civil; Hematologie Oncologie, Strasbourg
  - Hopitaux Du Leman Site Thonon; Maternite Gynecologie, Thonon-les-Bains
  - Clinique Pasteur; Oncologie Medicale, Toulouse
  - Clinique Saint Jean Languedoc; Oncologie Medicale, Toulouse
  - Hopital Bretonneau; Clinique D'Oncologie & de Radiotherapie, Tours
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
  - Hopital Prive Villeneuve d Ascq;Chimiotherapie Radiotherapie, Villeneuve-d'Ascq